CLINICAL TRIAL: NCT03902223
Title: A Randomized Screening Trial for Cardiac Sarcoidosis (CS) in Patients Seen During Routine Clinical Care Who Have Not Been Clinically Suspected to Have (CS), Comparing the Addition of Echocardiogram and Ambulatory ECG to Standard of Care.
Brief Title: Routine Cardiac Screening in Sarcoidosis Patients
Acronym: PAPLAND
Status: Completed | Type: Observational
Sponsor: Foundation for Sarcoidosis Research (Other)
Responsible Party: Sponsor
Other Study IDs: CSN504-002
Record Dates: First submitted 2019-03-25; First posted 2019-04-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sarcoidosis; Cardiac Sarcoidosis; Boeck's Disease; Besnier-Boeck Disease
Keywords: sarcoidosis; cardiac sarcoidosis; cardiac sarcoidosis screening
MeSH Terms: conditions — Sarcoidosis | interventions — Echocardiography; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Enhanced Screening Protocol For Cardiac Sarcoidosis: Arm will be randomly assigned to undergo enhanced screening methods (ambulatory ECG and echocardiogram) at month 0 and month 24, as well as a phone call/chart review at month 12.
  Interventions: Diagnostic Test: Enhanced Screening Protocol for Cardiac Sarcoidosis.
- Routine Screening for Suspected Cardiac Sarcoidosis: Arm will be randomly assigned for the routine standard of care/no intervention with enhanced screening methods. They will be offered the EKG and symptom check at months 0 and 24, as well as a phone call/chart review at month 12.
  Interventions: Diagnostic Test: Routine Screening for Suspected Cardiac Sarcoidosis

INTERVENTIONS:
Diagnostic Test: Enhanced Screening Protocol for Cardiac Sarcoidosis. — To utilize enhanced screening tests for cardiac sarcoidosis in an undiagnosed and potentially under-diagnosed patient population to determine the rate of missed cardiac sarcoidosis diagnosis. Following testing by the standard screening tests, this intervention includes a subsequent echocardiogram and a wearable ECG, also known as a Holter Monitor or ambulatory ECG.
  Other Names: Echocardiogram and ambulatory ECG
  Groups: Enhanced Screening Protocol For Cardiac Sarcoidosis
Diagnostic Test: Routine Screening for Suspected Cardiac Sarcoidosis — To utilize standard of care screening tests for cardiac sarcoidosis. This includes symptom check and a standard ECG.
  Other Names: Symptom check and standard ECG.
  Groups: Routine Screening for Suspected Cardiac Sarcoidosis

SUMMARY:
This protocol is an unblended randomized screening trial will have consecutive patients with no suggestion of cardiac sarcoidosis according to usual screening enroll in an enhanced screening protocol. The routine clinical care is to gather patient's history of symptoms and under go an ECG. If a patient has an abnormal results in standard screening, they typically have further evaluations as part of their routine medical care. These tests might include an echocardiogram, ambulatory ECG, and advanced cardiac imaging (MRI, PET scan as per local practice). A patient that has normal results on standard screening will be randomly assigned to enhanced screening at each center. Half the patients will be randomized to usual follow-up (annual symptom assessment and ECG) and the other half will be assigned to the enhanced screening (echocardiogram and ambulatory ECG at enrollment and at 24 months).

The investigators hypothesize that screening using conventional history, physical and ECG in the general sarcoidosis population, followed by appropriate advanced imaging testing, will result in the identification of a higher percentage of ascertained cardiac sarcoidosis than has been reported historically (2-5%). The investigators hypothesize that routine use of echocardiogram with strain and ambulatory ECG will identify additional patients who will have advanced imaging abnormalities or who meet criteria for cardiac sarcoidosis. The investigators further hypothesize that re-screening patients after 24 months with repeat echocardiogram and ambulatory ECG will identify additional patients with suspicion for cardiac sarcoidosis who had no abnormalities on the standard screening tests.

DETAILED DESCRIPTION:
Cardiac involvement is among the most feared complications of sarcoidosis, and it is the second leading cause of death from sarcoidosis. Autopsy studies and serial imaging studies in patients without cardiac symptoms suggest that approximately 25% of U.S. sarcoidosis patients have evidence of cardiac involvement. 3 Major manifestations of cardiac sarcoidosis include conduction delays, dysrhythmias, and cardiomyopathy. Given the increased recognition of cardiac involvement, prompt screening and diagnosis of cardiac sarcoidosis has been emphasized as a key priority for sarcoidosis research. Screening for cardiac sarcoidosis conventionally has relied on symptoms and electrocardiogram. However, there are no validated screening instruments for symptom assessment, and the usefulness of individual components of the medical history (e.g. palpitations, chest pain, presyncope) has not been assessed. In one study, symptom assessment was found to be less than 50% sensitive for identification of individuals with abnormal cardiac imaging studies. ECG performed poorly, with less than 10% sensitivity. Holter monitoring and echocardiogram were more sensitive than ECG in that study, identifying 50% and 25%, respectively, of those with imaging findings suggesting cardiac sarcoidosis (CS). The intensity of screening for CS in unselected sarcoidosis patients is controversial. The Heart Rhythm Society working group could not agree that echocardiogram or ambulatory ECG added significantly to conventional testing of eliciting cardiac symptoms and ECG; therefore, the working group was unable to recommend adding these procedures as a routine for all sarcoidosis patients. In a large series of Greek non-cardiac sarcoidosis patients, echocardiogram and ambulatory ECG added little prognostic information to usual care. On the other hand, more sophisticated echocardiographic techniques such as speckle tracking seem to provide independent prognostic information. In a second study, Holter monitoring and echocardiography abnormalities were both more common in those with MRI findings consistent with CS, although the usefulness of the tests disappeared in multivariable analysis. While history and ECG are considered the standard of care at present, there is a continuing need to identify markers of poor outcomes. Cardiac MRI and/or cardiac FDG-PET scan can identify large proportions of individuals with asymptomatic imaging abnormalities, but these scans are expensive, require specialized expertise to interpret, require radiation (PET scan) and are likely impractical for widespread use in all sarcoidosis patients. A second unresolved issue concerning screening for cardiac sarcoidosis is the frequency of re-screening sarcoidosis patients who demonstrate no evidence for cardiac sarcoidosis on an initial screen. The investigators hypothesize that screening using conventional history, physical and ECG in the general sarcoidosis population, followed by appropriate advanced imaging testing, will result in the identification of a higher percentage of ascertained cardiac sarcoidosis than has been reported historically (2-5%). The investigators hypothesize that routine use of echocardiogram with strain and ambulatory ECG will identify additional patients who will have advanced imaging abnormalities or who meet criteria for cardiac sarcoidosis. The investigators further hypothesize that re-screening patients after 24 months with repeat echocardiogram and ambulatory ECG will identify additional patients with suspicion for cardiac sarcoidosis who had no abnormalities on the initial screening tests.

Aims

1. To evaluate the rate of diagnosis of cardiac sarcoidosis during standard of care clinical practice that relies on patient symptoms and ECG.
2. To evaluate whether second-tier screening tests (echocardiogram and ambulatory ECG) improve the rate of diagnosis of cardiac sarcoidosis beyond conventional screening methods.
3. To evaluate the rate of diagnosis of cardiac sarcoidosis in sarcoidosis patients who had initial negative conventional and second-tier screening tests after undergoing these screening tests again at two years.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sarcoidosis as per The American Thoracic Society guidelines
2. First visit to the enrolling center
3. Intent to continue care at the enrolling center at least annually

Exclusion Criteria:

1. Referred to the enrolling center to evaluate for suspected cardiac sarcoidosis.
2. Pre-existing high suspicion for cardiac sarcoidosis, defined as having had cardiac MRI or cardiac PET scan, even if it was ordered by other institutions.
3. Severe sarcoidosis or other disease conferring a high likelihood of death or transplant within the next year
4. Unwilling or unable to undergo echocardiography and ambulatory ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with both suspected sarcoidosis and confirmed diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Positive result found from enhanced cardiac sarcoidosis screening at initial visit (sensitivity) | Day 1
  To evaluate whether second-tier screening tests (echocardiogram and ambulatory ECG) improve the rate of diagnosis of cardiac sarcoidosis beyond conventional screening methods.
Positive result found on enhanced cardiac screening at month 12 (sensitivity) | Month 12
  To evaluate whether second-tier screening tests (echocardiogram and ambulatory ECG) improve the rate of diagnosis of cardiac sarcoidosis beyond conventional screening methods during chart review.
Positive result found from enhanced cardiac screening at month 24 (sensitivity) | Month 24
  To evaluate the rate of diagnosis of cardiac sarcoidosis in sarcoidosis patients who had initial negative conventional and second-tier screening tests after undergoing these screening tests again at two years

SECONDARY OUTCOMES:
Positive result from study cohort | Up to 120 months after study completion
  To evaluate the rate of diagnosis of cardiac sarcoidosis in study cohort after 10 years.
Rate of diagnosis of cardiac sarcoidosis during standard of care of patient symptoms and ECG. | Up to 24 months from day 1
  To evaluate the rate of diagnosis of cardiac sarcoidosis during standard of care clinical practice that relies on patient symptoms and ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Culver, DO, Principal Investigator — The Cleveland Clinic; Muhunthan Thillai, MBBS, Principal Investigator — Royal Papworth Hospital
Locations (12):
- United States (10):
  - National Jewish Health, Denver, Colorado
  - Northwestern University Medicine, Chicago, Illinois
  - University of Illinois Medical Center At Chicago, Chicago, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Albany Medical Center, Albany, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington Medical Center, Seattle, Washington
- St. Antonius, Amsterdam, Nieuwegein, Netherlands
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be housed in a secured RedCap database. Protected health information (PHI) will be available only to the individual institutions, and the RedCap database will not house such data.
  Each subject will be entered into the database using a unique subject identifying number.